CLINICAL TRIAL: NCT05736328
Title: Effect of Lower Extremity Traction on the Popliteal Angle After Percutaneous Needle Tenotomy of the Knee Flexor Muscles.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de Sante Parasport Connecte Synergies (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-002
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Disability or Chronic Disease Leading to Disablement
Keywords: Neuro-Orthopaedics; Traction; Tenotomy; Disabled persons
MeSH Terms: interventions — Traction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects admitted for percutaneous needle tenotomy of the knee flexor muscles: Postoperative lower extremity traction.
  Interventions: Procedure: Traction

INTERVENTIONS:
Procedure: Traction — Postoperative lower extremity traction

SUMMARY:
People with neuromotor disability (i.e. following an inborn or acquired spinal cord, cerebral or peripheral neurological lesion) are at risk of neuro-orthopaedic disorders. Microinvasive percutaneous needle tenotomy is a frequent use alternative to open surgery to treat limb deformities. A lower extremity traction is performed in our unit during 2 to 7 days after surgery of the knee flexor muscles.

The aim of this study is to describe the efficiency of lower extremity traction on the popliteal angle after percutaneous needle tenotomy of the knee flexor muscles.

DETAILED DESCRIPTION:
This is a prospective, monocentric, cohort study of neurological disabled inpatients subjects treated in the perioperative disability unit (UPOH) of our university hospital for limb deformities by percutaneous needle tenotomy of the knee flexor muscles.

All eligible inpatient subjects with neuromotor disability and admitted for the treatment of limb deformities by percutaneous needle tenotomy of the knee flexor muscles will be consecutively included.

Data will be collected from the patients' medical records, in particular data related to their clinical, radiological, biological, and physiological examinations.

This is a routine care study; no procedures are added for research purposes. It is an ancillary study to the NO-AGING study.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old ;
* Treated in the Perioperative Disability Unit (UPOH) of the Physical Medicine and Rehabilitation Department of our university hospital;
* Admitted for the treatment of limb deformities by percutaneous needle tenotomy of the knee flexor muscles ;
* Having a neuromotor disability;
* No opposition to be enrolled in the study from the patient, or from a legally authorized close relative if the patient's state of health does not allow it;
* Affiliation to a social security scheme.

Exclusion Criteria:

* Associated open surgery ;
* Associated bone surgery ;
* Under court protection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with neuromotor disability and admitted for the treatment of limb deformities by percutaneous needle tenotomy of the knee flexor muscles.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Popliteal angle at the end of the traction | Daily, during the traction (up to 7 days).
  Difference in popliteal angle between the beginning and end of traction, evaluated with the Kinovea angle measurement tool. In case of bilateral traction, the average of the differences of each limb will be considered.

SECONDARY OUTCOMES:
Success of surgery | At 30 days after surgery
  Evaluated by the Goal Assessment Scale (GAS). Minimum and maximum values : -2 (worse outcome) / +2 (better outcome)
Popliteal angle | Daily, during the traction (up to 7 days).
  Evaluated by goniometry or Kinovea
Knee angle | Daily, during the traction (up to 7 days).
  Evaluated by goniometry or Kinovea
Pain | Daily, during the traction (up to 7 days).
  Numeric scale or Algoplus according to disability. Minimum and maximum values for the Numeric scale : 0 (no pain) / 10 (worst pain). Minimum and maximum values for the Algoplus scale : 0 (no pain) / 5 (worst pain).
Skin condition | Daily, during the traction (up to 7 days).
  Presence of erythema, phlyctens or superficial pressure sores

CONTACTS AND LOCATIONS:
Overall Officials: François Genêt, MD-PhD, Study Chair — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France; Vincent T. Carpentier, MD-MSc, Study Director — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France
Locations (1):
- Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chesnel C, Genet F, Almangour W, Denormandie P, Parratte B, Schnitzler A. Effectiveness and Complications of Percutaneous Needle Tenotomy with a Large Needle for Muscle Contractures: A Cadaver Study. PLoS One. 2015 Dec 1;10(12):e0143495. doi: 10.1371/journal.pone.0143495. eCollection 2015. PMID 26624990
- [Background] Schnitzler A, Genet F, Diebold A, Mailhan L, Jourdan C, Denormandie P. Lengthening of knee flexor muscles by percutaneous needle tenotomy: Description of the technique and preliminary results. PLoS One. 2017 Nov 7;12(11):e0182062. doi: 10.1371/journal.pone.0182062. eCollection 2017. PMID 29112966
- [Background] Angioni F, Salga M, Denormandie P, Genet F, Haigh O, David R, Gatin L, Schnitzler A. Microinvasive percutaneous needle tenotomy, An alternative to open surgery to treat neurological foot deformities. Ann Phys Rehabil Med. 2023 Mar;66(2):101690. doi: 10.1016/j.rehab.2022.101690. Epub 2022 Nov 30. No abstract available. PMID 35843500